CLINICAL TRIAL: NCT03041558
Title: SafeCare+: Implementing & Evaluating Trauma-Informed, Evidence-Informed Interventions for Latino Families Experiencing Domestic Violence & Child Maltreatment
Brief Title: Evaluating Trauma-Informed, Evidence-Informed Interventions for Latino Families Experiencing Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: South Bay Community Services (Unknown); University of Southern California (Other); San Diego County Child Welfare Services (Unknown); University of Oklahoma (Other); Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Principal Investigator, Gregory Aarons, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20140475
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Interpersonal Relations
Keywords: healthy relationships; interpersonal relations; domestic violence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SafeCare+ (SC+) (Experimental): SafeCare intervention with the additional Healthy Relationships (HR) module
  Interventions: Behavioral: SafeCare+ (SC+)
- SafeCare (SC) (Active Comparator): SafeCare intervention as usual
  Interventions: Behavioral: SafeCare (SC)

INTERVENTIONS:
Behavioral: SafeCare+ (SC+) — SafeCare intervention with the additional Healthy Relationships (HR) module
  Arms: SafeCare+ (SC+)
Behavioral: SafeCare (SC) — SafeCare intervention as usual
  Arms: SafeCare (SC)

SUMMARY:
This project will evaluate the implementation and efficacy of a domestic violence intervention module for parents receiving child welfare home visitation services.

DETAILED DESCRIPTION:
The ultimate goal of this proposed project is the provision of culturally-relevant, trauma-informed services leading to a reduction of family violence, and a resultant increase in family stability, improved communication, and a healthy home environment for children in Latino families with co-occurring domestic violence (DV) and child abuse/neglect (CAN). The Administration for Children, Youth and Families (ACYF) funded project and evaluation will be layered onto the existing UC San Diego's NIH-funded R01 research (NIH R01 MH092950) on scale-up of SafeCare (SC) across the entire San Diego Child Welfare System. In the first phase of this project, the community and academic partners will collaborate to develop a detailed evaluation plan by collecting formative qualitative data via focus groups with active CW clients with domestic violence (DV) histories and community child welfare and DV service providers. The second phase of this project will begin with the implementation of SafeCare+ (SC+), an evidence-based training curriculum for parents referred for child maltreatment, coupled with the Healthy Relationships (HR) module for Latino families with co-occurring child maltreatment and domestic violence experiences. SafeCare® (SC) has been shown to be widely accepted among the Latino community and the HR module has been specifically adapted for and successfully utilized with Latino populations. As part of the expansion of the original research study, 80 clients who will be recruited into the existing study will also be randomly assigned to receive the additional HR module.

ELIGIBILITY:
Inclusion Criteria:

* Service providers (CWS and DV) and active CW clients with DV histories will be recruited via random selection to participate in focus groups during the planning year of the project.
* Latino families are eligible for the RCT based on the following criteria: (a) being identified as an appropriate family for SafeCare; and (b) by having at least one, qualifying DV experience, which will be determined during the baseline needs assessment.

Exclusion Criteria:

* A client will be excluded if he/she indicates to the service provider that they are unable to comprehend the written questionnaire and cannot obtain outside assistance in understanding and completing the questionnaire.
* Clients under the age of 18 will able be excluded because they cannot provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Fidelity | 4 years
  Fidelity monitoring will begin simultaneously with the implementation of SafeCare (SC®). Fidelity is assessed largely via client report, with clients completing a fidelity questionnaire at the end of every SC or SC+ session. A secondary fidelity component utilizes information gained from the natural implementation of SC®. SC+ includes ongoing consultation in the form of expert SC® clinicians who accompany home visitors, observe their interactions with families, and coach them on improving performance and services.
Change in level of domestic violence | 4 years
  The Conflict Tactic Scale (CTS2): measures both the extent to which partners in a dating, cohabiting, or marital relationship engage in psychological and physical attacks on each other and also their use of reasoning or negotiation to deal with conflicts.
Client depression | 4 years
  The Center for Epidemiologic Studies Depression Scale (CES-D) (Radloff, 1977) is a 20-item questionnaire which assesses depressive symptomology.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fettes DL, Aarons GA, Brew V, Ledesma K, Silovsky J. Implementation of a trauma-informed, evidence-informed intervention for Latinx families experiencing interpersonal violence and child maltreatment: protocol for a pilot randomized control trial of SafeCare+(R). Pilot Feasibility Stud. 2020 Oct 8;6:153. doi: 10.1186/s40814-020-00681-3. eCollection 2020. PMID 33062294